CLINICAL TRIAL: NCT03297918
Title: Impact of a Structural Phonation Training on Respiratory Muscle Function in Patients With Structural Heart Disease - HeartChoir
Brief Title: Impact of a Structural Phonation Training on Respiratory Muscle Function in Patients With Structural Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HeartChoir
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure; Congenital Heart Disease
MeSH Terms: conditions — Heart Failure; Heart Defects, Congenital | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Interventional, single-center, randomised clinical trial
Who Masked: Participant
Masking Description: randomised
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Patients will be asked to participate in a structured singing and respiratory training for 12 weeks.
  Interventions: Behavioral: Respiratory muscle training
- Control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Respiratory muscle training — The intervention is two-parted and includes weekly singing lessons in a choir, held by a professional instructor, with additional instructions for daily breathing exercise at home.
  Arms: Intervention group

SUMMARY:
Most patients with complex congenital heart disease and cardiomyopathy from acquired heart disease have reduced exercise capacity. Exercise capacity is associated with respiratory muscle strength and function. If structured respiratory muscle training positively influences respiratory muscle function in patients with structural heart disease is not well known. The aim of this study is to investigate whether regular singing lessons and breathing exercises improve respiratory muscle strength in patients with congenital or acquired structural heart disease.

DETAILED DESCRIPTION:
Most patients with complex congenital heart disease and cardiomyopathy from acquired heart disease have reduced exercise capacity (VO2 max). Furthermore, exercise capacity is associated with respiratory muscle strength and function (maximal inspiratory (MIP) and maximal respiratory (MEP) pressures. If structured respiratory muscle training positively influences respiratory muscle function in patients with complex congenital heart disease or cardiomyopathy from acquired heart disease is not well known.

Aim: The aim of this study is to investigate the influence of a structured phonation and respiratory training with regular singing lessons on respiratory muscle strength and function (MIP and MEP), exercise capacity (VO2 max), NT-proBNP and quality of life.

This is an interventional, single-centre, randomized study. Patients will be recruited from the heart failure and congenital heart disease clinic of the University hospital Basel. Patients will be asked to participate in a structured phonation and respiratory muscle training for 12 weeks. The structured phonation and respiratory muscle training includes weekly singing lessons in a choir, held by a professional instructor, with additional instructions for daily respiratory muscle strength training at home. Respiratory muscle function (MIP and MEP), exercise capacity (VO2max) and quality of life will be measured at the beginning of the intervention and after 12 weeks of interventional training. In parallel, respiratory muscle function, exercise capacity, NT-proBNP and quality of life will be measured in a gender and age matched group of patients without performing the intervention and in a healthy control group who co-participate the choir lessons and the respiratory muscle training. Primary endpoint is the change of maximal inspiratory pressures (MIP) between patients with and without a structured phonation and respiratory muscle training. Secondary endpoints are changes of MEP, VO2max, NT-proBNP and quality of life between patients with and without the intervention; changes of all measured variables between patients and the healthy control group, and changes of all measured variables before and after the intervention in patients. Inclusion criteria: Patients >18 years with known cardiomyopathy from acquired heart disease (ischemic or dilated) or complex forms of congenital heart disease. Exclusion criteria: Acute coronary syndrome ≤6 months or heart failure hospitalization ≤12 months.

Structural singing lesions and respiratory muscle function training may improve respiratory muscle strength, exercise capacity and quality of life in patients with heart failure or complex congenital heart disease. The intervention comes at low costs, can be applied by most of the patients and is feasible even for disabled patients who are not able to participate in regular exercise training. Furthermore, singing may improve respiratory muscle strength and exercise capacity even in the healthy population.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* age ≥ 18 years
* known cardiomyopathy from acquired heart disease (ischemic or dilated) or patients with complex CHD (cyanotic congenital heart disease, Fontan palliation, subaortic right ventricle or repaired tetralogy of Fallot)

Exclusion Criteria:

* Acute coronary syndrome, cardiac surgery or heart failure hospitalization within the previous 6 months
* chronic metabolic, orthopedic, or infectious disease; treatment with steroids, hormones, or cancer chemotherapy
* severe exercise-induced asthma
* professional singer or professionally performing a wind instrument
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure in kilopascal | 12 weeks
  Change of maximal inspiratory pressure after the intervention

SECONDARY OUTCOMES:
Change of MEP | 12 wees
  Change of maximal expiratory pressure after the intervention
Change of MVO2 | 12 weeks
  Change of maximal VO2 after the intervention
Change of QoL | 12 weeks
  Change of Quality of life
NT-proBNP | 12 weeks
  Change of Level of NT-proBNP after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tobler, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ganzoni C, Arslani K, Pfister O, Freese M, Strobel W, Mueller C, Tobler D. Choir singing improves respiratory muscle strength and quality of life in patients with structural heart disease - HeartChoir: a randomised clinical trial. Swiss Med Wkly. 2020 Sep 16;150:w20346. doi: 10.4414/smw.2020.20346. eCollection 2020 Sep 7. PMID 33038262